CLINICAL TRIAL: NCT06725615
Title: Umami Exposure on MSG-induced Satiation
Brief Title: Effect of Umami Exposure on MSG Induced-satiation
Acronym: RISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Ciaran Forde, Prof. Dr., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL88298.091.24
Record Dates: First submitted 2024-11-27; First posted 2024-12-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Sensory Testing; Umami Taste Perception; Food Intake Regulation
Keywords: umami; taste; intensity; ad libitum; intake; exposure

STUDY DESIGN:
Intervention Model Description: Randomised controlled intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Regular Umami exposure (Experimental): The Regular Umami Exposure (RegularU) group (control) will receive the basic diet with added MSG, representing Dutch dietary intake levels of around the 50th percentile, which is about 20-25 mg/kg body weight.
  Interventions: Other: Regular Umami exposure; Other: one-week run-in period
- High Umami exposure (Experimental): the High Umami Exposure (HighU) will receive the basic diet with added MSG, representing Dutch intake levels of around the 90th percentile, which is about 50-55 mg/kg body weight.
  Interventions: Other: High Umami exposure; Other: one-week run-in period
- Low Umami exposure (Experimental): The Low Umami Exposure (LowU) group will receive the basic diet without added MSG.
  Interventions: Other: Low Umami exposure; Other: one-week run-in period

INTERVENTIONS:
Other: Regular Umami exposure — This group will receive the basic diet with added MSG, representing Dutch intake levels of around the 50th percentile, which is about 20-25 mg/kg body weight.
  Arms: Regular Umami exposure
Other: High Umami exposure — This group will receive the basic diet with added MSG, representing Dutch intake levels of around the 90th percentile, which is about 50-55 mg/kg body weight.
  Other Names: HighU
  Arms: High Umami exposure
Other: Low Umami exposure — This group will receive the basic diet without added MSG.
  Other Names: LowU
  Arms: Low Umami exposure
Other: one-week run-in period — During the one-week run-in period, all participants will receive the RegularU diet, which is the basic diet with added MSG, representing Dutch intake levels of around the 50th percentile (about 20-25 mg MSG intake daily per kg body weight).
  Other Names: run-in

SUMMARY:
Monosodium Glutamate (MSG) is an amino acid salt that naturally enhances umami taste in many foods. It is often used to reduce salt (NaCl) in products while keeping the flavour. However, MSG might slow down satiation, leading to larger portions. This effect could vary based on diet and umami exposure, but there is no empirical data yet to confirm this hypothesis. Therefore, a long-term systematic investigation is necessary to objectively evaluate what the duration and extent of the effect of umami taste exposure is on absolute food intake, and whether it can have an effect on other outcomes, such as appetite ratings, meal liking, taste sensitivity, food preference, body hydration, weight status, self-reported diet tolerance and other potential side effects. The study sample will consist of 75 participants, that will randomly be distributed over three intervention groups: regular umami exposure (n = 25), low umami exposure (n = 25) and high umami exposure (n = 25). The intervention is fully controlled, for a period of two weeks, with an additional one-week run-in period in which all participants consume the regular umami exposure diet. Umami taste will be added through MSG supplementation of the three main meals. Supplementation will depend on both intervention group, and individual participants' body weight. The primary objective is to compare the effects of a 2-week low-, regular- and high dietary MSG exposure on umami-induced satiation. Differences in absolute food intake will be assessed by an ad libitum satiation test, which participants will be presented with at baseline (day 7), mid-intervention (day 14) and end of intervention (day 22). Secondary outcomes such as differences between intervention groups in satiety and appetite ratings, test meal liking, taste sensitivity, food preference, body hydration status, weight, self-reported diet tolerance and other potential side effects.

DETAILED DESCRIPTION:
Umami seems to have a dual role in food intake regulation. On the one hand, flavouring meals with MSG has been shown to increase meal size by enhanced palatability. On the other hand, it has also shown to decrease food intake on the longer term. For example, studies with MSG supplemented preloads report lower hunger ratings, desire to eat, or reduced food intake compared to a control. So, although MSG enhances the palatability of meals and increases initial meal sizes, it may be effective in reducing hunger and subsequent food intake later in the day. Therefore, long-term, studies isolating umami taste are needed, to be able to examine its duration and extent of effect on food intake. In the proposed study, we compare the effects of diets with different levels of umami taste on different aspects of energy intake regulation. It primarily aims to study the effect of dietary exposure to umami taste on umami-induced satiation; to answer questions on the effect size and direction, and duration of effects. The intervention approach - using population distribution of taste exposure - builds upon a study that we recently conducted on the effect of sweetness exposure on dietary behaviour, keeping the taste exposure within realistic boundaries and therefore relevant for the Dutch population. The study will provide important data on the health effects of MSG use in food reformulations within realistic boundaries; it will give insights in food intake regulation and weight management. It may also guide health councils and other authorities in establishing realistic dietary guidelines.

The primary objective is to compare the effects of a 2-week low, regular and high umami exposure on MSG-induced satiation. The hypothesis is that a low umami exposure will lead to a higher ad libitum food intake due to lower umami-induced satiation, and that a high umami exposure will lead to a lower ad libitum food intake in due to higher umami-induced satiation compared to regular umami exposure. Secondary objectives are to compare the effects of a 2-week low, regular and high umami exposure on satiety, appetite ratings, test food liking, taste sensitivity, food preference, body hydration status, weight status and self-reported MSG tolerance. Participants will be matched on sex (male or female), age (20-30 or 31-55) and weight (60-68kg, 68-77kg or 77-85kg) and randomly allocated to one of the three intervention arms:

* Low umami exposure, 0g MSG added to the diet daily (n = 25);
* Regular umami exposure (control), 20-25 mg MSG per kg body weight added to the diet daily (n = 25);
* High umami exposure, 50-55mg MSG per kg body weight added to the diet daily (n = 25).

The umami exposure level of the intervention diets is based on the estimated distribution of free glutamate intake of the Dutch population. The low umami intervention group represents 0-5% of the intake level, the regular umami intervention group represents 45-55% of the intake level, and the high umami intervention group represents 85-95% of the intake level. The intervention is fully controlled, meaning that participants will only consume foods they will be provided with for three weeks. Foods will be prepared and packed for participants individually, matching their energy needs, meaning that participants are required to consume everything they are provided with. A basic diet will be made, as low in naturally occurring free glutamate as possible, and supplemented with MSG according to participants' intervention group and body weight. Macronutrient composition of the offered foods is similar in energy and macronutrient composition, that is fat, protein, carbohydrates and fibers, but different in MSG content. To account for differences in sodium content, diets are matched using salt (NaCl) to ensure similar sodium intake. To account for baseline differences in umami tasting food intake, a one-week run-in period precedes the two-week dietary intervention. During this week, participants consume the regular umami exposure diet (control), as it allows for adjusting the energy provided by the diet. More importantly, it helps participants to get used to the diet, and it ensures that the three intervention groups start with the same baseline umami exposure.

MSG induced satiation will be assessed by measuring absolute food intake from an ad libitum containing meal. The main outcome is the difference in intake between intervention groups at the end of the intervention (day 22), adjusted for baseline differences (day 7). This is calculated as the mean intake at day 22 minus the intake at day 7 in both weight (g) and energy (kcal) per intervention arm. A mid-intervention measurement will be done on day 14, to assess a possible pattern of MSG induced satiation. Differences between intervention groups in satiety and appetite ratings and test meal liking will be assessed using a visual analogue scale in a short questionnaire daily and more elaborately on day 7, 14 and 22. Taste sensitivity, food preference, body hydration status and weight status will be measured on day 7, 14 and 22. Self-reported diet tolerance and other potential side effects will be measured daily in the participant's diary. Compliance will be assured by visiting the research facilities for lunch daily on weekdays, and by before and after lunch meal pictures during weekends.

ELIGIBILITY:
Inclusion Criteria:

* Healthy: as judged by the participant
* Age 20-55 years at the time of inclusion, assessed by date of birth;
* Proper understanding of the Dutch language, as questionnaires will be in Dutch;
* Able to visit Wageningen University, as required for dietary intervention and testing;
* Weight 60-80 kg (female) or 65-85 kg (male), as MSG supplementation is based on bodyweight;
* Body mass index 20-25 kg/m2;
* Having normal taste ability, assessed using Mueller taste strip test, ≥12 out of 20 assessed correctly;
* Able to provide informed consent.

Exclusion Criteria:

* Suffering from endocrine- or gastro-intestinal diseases or other diseases that might influence study outcomes (such as diabetes, Crohn's disease, cardiovascular disease, hypertension, etc.);
* Diagnosed with eating disorders (in the past);
* Diagnosed with taste or smell disorders in the past six months;
* Pregnant or lactating during the study intervention;
* Gain or loss of more than 3 kgs in the last three months prior to study entry;
* Suffering from lack of appetite for any reason;
* Use of medication that may influence the appetite, or medication that may affect body hydration status (medication will be judged by the medical investigator);
* Having a food allergy and/or intolerance for foods used in the dietary intervention (e.g. lactose intolerance, gluten intolerance, MSG sensitivity). This will be assessed with an open question;
* Consumes more than 14 (women) or 21 (men) glasses of alcohol per week;
* Consumes MSG-rich sauces (soy sauce, ketchup and/or curry paste) more than once per day, or consumes more than 3 savoury food items (paprika chips, instant noodles, sundried tomatoes and/or mushrooms) per day. This will be assessed with a frequency of consumption table;
* Irregular eating pattern. This will be measured with a frequency of meal/food consumption table, and is defined as: frequency of breakfast consumption less than once per week;
* Unwilling to maintain regular exercise pattern during the study period. This will be assessed with a yes/no question;
* Unwilling to quit use of soft or hard drugs during the intervention;
* Student or personnel of the division of Human Nutrition and Health, Wageningen University;
* Participating in any other intervention study/studies or planning to participate in another intervention study during the study period;
* Restrained eating score of ≥2.7 (females)/ ≥2.2 (males) measured by Dutch Eating Behaviour Questionnaire.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
MSG-induced satiation | From baseline to end of intervention (day 7 to day 22).
  The main outcome is the difference in intake between intervention groups at day 22, adjusted for baseline differences at day 7. This is calculated as the mean intake at day 22 minus the mean intake at day 7, in energy (kcal), per intervention arm. A mid-intervention measurement will be done on day 14.

SECONDARY OUTCOMES:
Changes in appetite and thirst ratings | From baseline to end of intervention (day 7 to day 22).
  The difference in appetite and thirst ratings between intervention groups at day 22, adjusted for baseline differences at day 7. This measure will be taken daily before the intervention meal, and three times (before, immediately after, and two hours after) around the ad libitum test meal. The questionnaire will consist of 6 questions, which will be rated on a visual analogue scale (0, not at all to 100 a lot).
Changes in liking of the ad libitum test meal | From baseline to end of intervention (day 7 to day 22).
  The difference in test meal liking between intervention groups at day 22, adjusted for baseline differences at day 7. A mid intervention measure will be done on day 14. This measure will be taken three times (before, immediately after, and two hours after) around the ad libitum test meal. The questionnaire will consist of 6 questions, which will be rated on a visual analogue scale (0, not at all to 100 a lot).
Changes in food preference | From baseline to end of intervention (day 7 to day 22).
  The difference in food preference between intervention groups at day 22, adjusted for baseline differences at day 7. Food preference will be measured by the Macronutrient and Taste Preference Ranking Task (MTPRT), which will be filled in on day 7, 14 and 22.
Changes in taste sensitivity | From baseline to end of intervention (day 7 to day 22).
  The difference in taste sensitivity between intervention groups at day 22, adjusted for baseline differences at day 7. Taste sensitivity will be assessed using the Mueller Taste Strip test, on day 7, 14 and 22.
Changes in body hydration status | From baseline to end of intervention (day 7 to day 22).
  The difference in body hydration status between intervention groups at day 22, adjusted for baseline differences at day 7. Body hydration status will be measured by freezing a spot-urine sample, and urine osmolality will be assessed, on day 7, 14 and 22.
Changes in Waist to hip ratio | From baseline to end of intervention (day 7 to day 22).
  The difference in body composition between intervention groups at day 22, adjusted for baseline differences at day 7. Body composition will be measured by waist-hip ratio using a stretch resistant tape, on day 7, 14 and 22.
Difference in bodyweight | Screening and day 1, 3, 7, 10, 14, 17, 22
  The difference in bodyweight between intervention groups at day 22, adjusted for baseline differences at day 7. Bodyweight will be measured by a weighing on a calibrated scale without sweater, belt or shoes, on day 7, 14 and 22. The average of two measures will be taken, and rounded to the closest decimal.
Difference in Adverse events occurence, or medication use | From start to end of intervention (day 1 to day 22).
  The difference in Adverse events occurence, or medication use between intervention groups at day 22, adjusted for baseline differences at day 7. This will be measured daily by a questionnaire in the study diary.
Weekend meal consumption | Start to end of study (day 1 to day 22), on weekend days
  Weekend meal consumption will be measured by assessing before and after pictures of weekend meals. This is a compliance measure, and will be done six times in total (3 weekends during the intervention, so 6 weekend days).
Changes in time effects of MSG-induced satiation | From baseline to mid of intervention (day 7 to day 14), and from mid of intervention to end of intervention (day 14 to day 21).
  This is defined as the difference in intake between intervention groups at mid-intervention (day 14), adjusted for baseline differences at day 7, and the difference in intake between intervention groups at end of intervention (day22) adjusted for mid-intervention differences at day 14. This is calculated as the mean intake at day 14 minus the mean intake at day 7, as well as the mean intake at day 22 minus the mean intake at day 14 in energy (kcal), in all three intervention arms. This mid-intervention measurement of MSG induced satiation will be done to assess possible time effects.

OTHER OUTCOMES:
Gender | Baseline (day 0)
  Based on self-report in the screening questionnaire. Baseline characteristic.
Age | Baseline (day 0)
  Based on self-report in the screening questionnaire. Baseline characteristic.
Height | Baseline (day 0)
  Will be assessed using a stadiometer as the average of two measurements, rounded to the closest decimal. This will be done during the physical screening session.
Baseline medicine usage | Baseline (day 0)
  Based on self-report in the screening questionnaire. Baseline characteristic.
Smoking status | Baseline (day 0)
  Based on self-report in the screening questionnaire. Baseline characteristic.
Dietary restraint score | Baseline (day 0)
  Measured by Dutch Eating Behaviour Questionnaire (DEBQ). This is an exclusion criterium: Restrained eating score of ≥2.7 (females)/ ≥2.2 (males) (scores range from 1-5).
Baseline savoury food consumption | Day 1 of the intervention
  Measured by Food Frequency Questionnaire designed to classify people on taste consumption patterns (tasteFFQ). Results will be used to describe the baseline consumption of savoury foods among test participants.
Habitual energy consumption | Screening (day 0)
  Measured by Food Frequency Questionnaire (FFQ), to be able to group participants on their energy needs, and to assign the correct amount of energy daily during the intervention.
Physical activity level | Screening and day 7, 14 and 22 of intervention
  Measured using the SQUASH questionnaire with a reference period of one week. This is a compliance measure as participants are asked to maintain stable exercise patterns during the study period. Physical activity will be reported as a along with descriptive measures of participant characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in an article after de-identification will be shared.
Supporting Information: SAP, Analytic Code
Time Frame: Following the publication. No end date.
Access Criteria: Anyone who whishes to access the data for secondary analysis must contact corresponding authors of specific publications for their approval. Next to this, they must reference the source of the data to provide appropriate credit to those who generated the data and allow searching for the studies it has supported.

REFERENCES:
- [Background] Terpstra SES, Hoogervorst LA, van der Velde JHPM, Mutsert R, van de Stadt LA, Rosendaal FR, Kloppenburg M. Validation of the SQUASH physical activity questionnaire using accelerometry: The NEO study. Osteoarthr Cartil Open. 2024 Mar 18;6(2):100462. doi: 10.1016/j.ocarto.2024.100462. eCollection 2024 Jun. PMID 38577551
- [Background] Geha RS, Beiser A, Ren C, Patterson R, Greenberger PA, Grammer LC, Ditto AM, Harris KE, Shaughnessy MA, Yarnold PR, Corren J, Saxon A. Review of alleged reaction to monosodium glutamate and outcome of a multicenter double-blind placebo-controlled study. J Nutr. 2000 Apr;130(4S Suppl):1058S-62S. doi: 10.1093/jn/130.4.1058S. PMID 10736382
- [Background] Cad EM, Tang CS, de Jong HBT, Mars M, Appleton KM, de Graaf K. Study protocol of the sweet tooth study, randomized controlled trial with partial food provision on the effect of low, regular and high dietary sweetness exposure on sweetness preferences in Dutch adults. BMC Public Health. 2023 Jan 11;23(1):77. doi: 10.1186/s12889-022-14946-4. PMID 36627602
- [Background] Imada T, Hao SS, Torii K, Kimura E. Supplementing chicken broth with monosodium glutamate reduces energy intake from high fat and sweet snacks in middle-aged healthy women. Appetite. 2014 Aug;79:158-65. doi: 10.1016/j.appet.2014.04.011. Epub 2014 Apr 23. PMID 24768895
- [Background] Anderson GH, Fabek H, Akilen R, Chatterjee D, Kubant R. Acute effects of monosodium glutamate addition to whey protein on appetite, food intake, blood glucose, insulin and gut hormones in healthy young men. Appetite. 2018 Jan 1;120:92-99. doi: 10.1016/j.appet.2017.08.020. Epub 2017 Aug 24. PMID 28843973
- [Background] van Avesaat M, Troost FJ, Ripken D, Peters J, Hendriks HF, Masclee AA. Intraduodenal infusion of a combination of tastants decreases food intake in humans. Am J Clin Nutr. 2015 Oct;102(4):729-35. doi: 10.3945/ajcn.115.113266. Epub 2015 Aug 19. PMID 26289437
- [Background] Masic U, Yeomans MR. Does monosodium glutamate interact with macronutrient composition to influence subsequent appetite? Physiol Behav. 2013 May 27;116-117:23-9. doi: 10.1016/j.physbeh.2013.03.017. Epub 2013 Mar 24. PMID 23531472
- [Background] Masic U, Yeomans MR. Umami flavor enhances appetite but also increases satiety. Am J Clin Nutr. 2014 Aug;100(2):532-8. doi: 10.3945/ajcn.113.080929. Epub 2014 Jun 18. PMID 24944058
- [Background] Bellisle F, Monneuse MO, Chabert M, Larue-Achagiotis C, Lanteaume MT, Louis-Sylvestre J. Monosodium glutamate as a palatability enhancer in the European diet. Physiol Behav. 1991 May;49(5):869-73. doi: 10.1016/0031-9384(91)90196-u. PMID 1886949